CLINICAL TRIAL: NCT07164560
Title: Clinical Study of TRBC1/2-Targeted CAR-T Cells in the Treatment of Relapsed/Refractory Peripheral T-Cell Lymphoma
Brief Title: Exploratory Study of TRBC1/2-Targeted CAR-T Cell Therapy in Relapsed/Refractory Peripheral T-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0638
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Refractory/Recurrent Peripheral T-cell Lymphoma
Keywords: Refractory/recurrent; TRBC1/2 CAR-T; Peripheral T-cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PB TRBC1/2 CAR-T (Experimental)
  Interventions: Biological: Anti-TRBC1 CAR-T cells

INTERVENTIONS:
Biological: Anti-TRBC1 CAR-T cells — lentiviral vector-transducted peripheral blood-derived T cells to express anti-TRBC1 CAR

SUMMARY:
This study aims to evaluate the safety and efficacy of TRBC1/2-directed chimeric antigen receptor T cells (TRBC1/2 CAR-T cells) in patients with refractory or relapsed peripheral T-cell lymphoma (PTCL).

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, phase I clinical trial designed to evaluate the safety and efficacy of TRBC1/2 CAR-T cell therapy in patients with TRBC1/2-positive T-cell lymphoma.

The study will be conducted in two parts:

Phase I (Dose Escalation):

A dose-escalation study will be carried out following the conventional "3+3" design, with one dose level administered via intravenous infusion. Each cohort will enroll 3 to 6 patients. After the initial infusion, patients will be observed for at least 28 days for safety evaluation, followed by long-term follow-up of up to 2 years post-infusion.

Phase II (Dose Expansion):

Based on safety, in vivo expansion and persistence of TRBC1/2 CAR-T cells, and preliminary efficacy results from Phase I, the recommended dose and administration schedule will be determined. Approximately 30 eligible patients will then be enrolled to further assess safety and efficacy at the selected dose. Following the first infusion of TRBC1/2 CAR-T cells, patients will continue in long-term follow-up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria

According to the 2016 WHO classification of lymphoid neoplasms, patients with relapsed/refractory peripheral T-cell lymphoma (PTCL) must meet the following criteria to be eligible for enrollment:

1. Voluntarily agree to participate in this study and provide signed informed consent.
2. Age 18 to 75 years, male or female.
3. Diagnosis of relapsed/refractory PTCL, defined as failure of ≥1 prior line of therapy. Eligible histologic subtypes include (but are not limited to):

   Angioimmunoblastic T-cell lymphoma (AITL) Anaplastic large cell lymphoma (ALCL) Peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS)
4. Estimated life expectancy ≥12 weeks.
5. TRBC1/2-positive tumor tissue (≥20% by immunohistochemistry) OR TCR gene rearrangement confirmed by PCR or NGS.
6. ECOG performance status of 0-2.
7. Adequate organ function as defined below:

   ALT and AST ≤ 2.5 × upper limit of normal (ULN) Creatinine clearance (Cockcroft-Gault) ≥ 60 mL/min Total bilirubin ≤ 1.5 × ULN Left ventricular ejection fraction (LVEF) ≥ 50% Baseline oxygen saturation > 92% on room air

   Hematology:

   Phase Ia: ANC > 1500/mm³, platelets > 75 × 10⁹/L, hemoglobin > 9 g/dL Phase Ib: ANC > 1000/mm³, platelets > 50 × 10⁹/L, hemoglobin > 8 g/dL
8. ≥3 months since prior autologous hematopoietic stem cell transplantation.
9. Prior CAR-T therapy targeting a different antigen is permitted if lack of efficacy was confirmed after ≥3 months of evaluation, or if complete remission (CR) was achieved but relapse occurred.
10. Women of childbearing potential must have a negative pregnancy test prior to enrollment. All patients (male and female) must agree to use effective contraception during the study.
11. Presence of at least one measurable lesion.
12. All approved prior anti-tumor therapies (including systemic chemotherapy, total body irradiation, or immunotherapy) must have been completed ≥3 weeks before study drug administration; for non-chemotherapy targeted agents, a washout period of ≥2 weeks is required.

Exclusion Criteria

Patients meeting any of the following criteria will be excluded from this study:

1. History of allergy to any component of the cell product.
2. History of another malignancy that has not achieved remission.
3. Prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
4. Receipt of gene therapy within the past 3 months.
5. Uncontrolled systemic active infection (with the exception of simple urinary tract infection or bacterial pharyngitis). Prophylactic use of antibiotics, antivirals, or antifungal agents is permitted.
6. Active hepatitis B infection (HBsAg positive; however, patients with HBV-DNA <10³ copies/mL are not excluded), active hepatitis C virus infection (including carriers), syphilis, or other acquired or congenital immunodeficiency diseases, including but not limited to HIV infection.
7. New York Heart Association (NYHA) Class III or IV heart failure.
8. Unresolved toxicity from prior anti-tumor therapy (defined as CTCAE v5.0 Grade >1, with the exception of fatigue, anorexia, and alopecia).
9. Evidence of central nervous system (CNS) involvement at screening, or clinically significant CNS disease such as a history of seizures or other CNS disorders.
10. Prior exposure to any agent specifically targeting TRBC1/2.
11. Lactating women who are unwilling to discontinue breastfeeding.
12. Any other condition that, in the opinion of the investigator, may increase patient risk or interfere with the study results.
13. Autoimmune disease requiring immunosuppressive therapy.
14. Use of immunosuppressive agents or therapeutic doses of corticosteroids (defined as prednisone >20 mg/day or equivalent) within 7 days prior to leukapheresis, or use of hematopoietic growth factors such as G-CSF. Physiological replacement therapy, topical, or inhaled corticosteroids are permitted.
15. Receipt of chemotherapy, targeted therapy, immunotherapy, or radiotherapy within 3 days prior to leukapheresis.
16. Participation in another clinical trial within 4 weeks or within 5 half-lives of the investigational product (whichever is shorter) prior to leukapheresis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of peripheral blood-derived Anti-TRBC1/2 CAR-T Cell Therapy for refractory/relapsed peripheral T-cell lymphoma.

SECONDARY OUTCOMES:
Complete response rate (CR) | 3 months
  To determine the anti-tumor effectivity of PB TRBC1/2 CAR-T

OTHER OUTCOMES:
Overall response rate (ORR) | 3 months
  To determine the anti-tumor effectivity of PB TRBC1/2 CAR-T
Progression free survival (PFS) | Up to 2 years
  To determine the anti-tumor effectivity of PB TRBC1/2 CAR-T
Overall survival (OS) | Up to 2 years
  To determine the anti-tumor effectivity of PB TRBC1/2 CAR-T
Duration of response (DOR) | Up to 2 years
  To determine the anti-tumor effectivity of PB TRBC1/2 CAR-T

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital,School of Medicine,Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No